CLINICAL TRIAL: NCT06228781
Title: Autologous Hematopoietic Stem Cell Transplantation for Refractory Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Qiang Liu, Professor of Department of Neurology, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB2023-YX-233-01
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): Patients will undergo stem cell transplantation for the treatment of refractory MS
  Interventions: Procedure: Autologous haemopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Autologous haemopoietic stem cell transplantation — Immuno-ablation and autologous CD34 selected hematopoietic stem cell transplantation (HSCT).
  Stem cell mobilization with cyclophosphamide 2g/m2 and filgrastim 10 ug/kg/d x 5 day.
  Stem cell collection with cobe cpectra stem cell purification with Miltenyi CliniMACS Stem cell transplant conditioning with busulphan 3.2 mg/kg ; fludarabine 30mg/m2 or cladribine 10mg ；cytarabine 1-2g/m2 or idarubicin 8mg/m2；cyclophosphamide 40mg/kg followed by CD34 selected autologous hematopoietic stem cell transplant.

SUMMARY:
Autologous hematopoietic stem cell transplantation (aHSCT) is the only treatment for refractory autoimmune diseases capable of inducing long-term, drug-free and asymptomatic remission. Over the past two decades, aHSCT has been used to treat inflammatory autoimmune disease of the CNS. Patients with relapsing-remitting multiple sclerosis benefit from aHSCT treatment. However, a certain percentage of patients still experience recurrence 3 or 5 years after transplantation. Therefore, exploration of conditioning regimens will drive therapeutic advances in aHSCT in autoimmune diseases of the CNS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years;
2. Diagnosed multiple sclerosis with relapses or progression and sustained accumulated impairment by a neurologist expert in the field;
3. EDSS score of 3-6 (including 3 and 6);
4. EDSS cerebellar functional score ≥ 3 or EDSS pyramidal functional score ≥3；
5. Evidence of current disease activity;
6. If a patient has previously received a cytotoxic agent (mitoxantrone, cyclophosphamide etc.) they must have normal bone marrow morphology and cytogenetics before being considered eligible for this study ;
7. No evidence of hepatic inflammation or fibrosis;

Exclusion Criteria:

1. Patients with evidence of myelodysplasia or other non-autoimmune cytopenia;
2. Patients having received a cytotoxic agent within one month of enrolling in this study;
3. Patient with any active or chronic infection (herpes simplex virus, varicella-zoster virus, cytomegalovirus, EB virus, human immunodeficiency virus, hepatitis virus, syphilis, etc.);
4. Patients having received a cytotoxic agent within one month of enrolling in this study;
5. Patients with a malignant tumor currently or within the last 5 years;
6. Patients with cardiac, renal, pulmonary, hepatic or other organ impairment;
7. Patients whose life expectancy is severely limited by another conditions;
8. Pregnancy or risk of pregnancy;
9. Patients unable to give written informed consent in accordance with research ethics board guidelines.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
3 year MS activity free survival | 3 year follow-up post transplant
  The events for the primary outcome are: clinical relapse, appearance of a new or Gd-enhancing lesion on MRI, or sustained progression of EDSS score.

SECONDARY OUTCOMES:
Time to MS treatment failure | 3 years
  Disease activity and disability will be assessed with clinical relapse, appearance of a new or Gd-enhancing lesion on MRI, or sustained progression of EDSS score and quality of life.
Transplant related morbidity | 3 years
  Rate of transplant related events.
Transplant related mortality | 3 years
  Rate of transplant related death.
Immune reconstitution following transplant | 3 years
  Rate of immune reconstitution following transplant.
Hematopoietic reconstitution following transplant | 3 years
  Rate of hematopoietic reconstitution following transplant.
Imaging changes associated with the disease activity | 3 years
  Imaging changes include:
  new or enlarging T2-weighted lesion count and new T1-weighted lesion count at all scans after baseline; T2-weighted lesion volume; Gd-enhanced lesion count and volume; and total volume of non-enhancing T1-weighted lesions on all MRI scans.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Liu, M.D.,Ph.D, Principal Investigator — Tianjin Medical University General Hospital